CLINICAL TRIAL: NCT04913012
Title: Sustainability of Exercise Therapy by the Use of Exercise Booster Sessions in People With Multiple Sclerosis.
Brief Title: Exercise Booster Sessions in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laurits_Madsen_PhD
Record Dates: First submitted 2021-05-26; First posted 2021-06-03 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Aerobic training booster group (Experimental): Will receive 12 weeks of aerobic training followed by booster sessions + standard care in the 40 follow up period
  Interventions: Combination Product: Systematic aerobic training; Combination Product: Aerobic training booster sessions
- Aerobic training control group (Active Comparator): Will receive 12 weeks of aerobic training followed by standard care in the 40 follow up period
  Interventions: Combination Product: Systematic aerobic training
- Resistance training booster group (Experimental): Will receive 12 weeks of resistance training training followed by booster sessions + standard care in the 40 follow up period
  Interventions: Combination Product: Systematic resistance training; Combination Product: Resistance training booster sessions
- Resistance training control group (Active Comparator): Will receive 12 weeks of resistance training followed by standard care in the 40 follow up period
  Interventions: Combination Product: Systematic resistance training
- Control group (No Intervention): Will receive standard care throughout the study

INTERVENTIONS:
Combination Product: Systematic aerobic training — Two-three weekly supervised aerobic exercise sessions for 12 weeks. The training will be planned by exercise physiologists, and performed in a progressive manner.
  Arms: Aerobic training booster group; Aerobic training control group
Combination Product: Systematic resistance training — Two-three weekly supervised resistance exercise sessions for 12 weeks. The training will be planned by exercise physiologists, and performed in a progressive manner.
  Arms: Resistance training booster group; Resistance training control group
Combination Product: Aerobic training booster sessions — Supervised aerobic training booster sessions delivered in the follow up period (two sessions every fifth week).
  Arms: Aerobic training booster group
Combination Product: Resistance training booster sessions — Supervised resistance training booster sessions in the follow up period (two sessions every fifth week).
  Arms: Resistance training booster group

SUMMARY:
This study wants to investigate whether exercise booster sessions applied in the follow-up period after an exercise intervention can increase the sustainability of exercise induced effects in persons with multiple sclerosis.

The study will be a randomized, multi-site, controlled trial. Participants will from the beginning be allocated to either aerobic training group, resistance training group or control group. After a 12 week exercise intervention, the exercise groups will be additionally randomized to receive either exercise booster sessions + standard care or just standard care in the 40 week follow up period.

It is hypothesized that exercise booster sessions can increase the sustainability of exercise induced effects.

DETAILED DESCRIPTION:
MS is a chronic, autoimmune, and inflammatory disease of the central nervous system, exemplified through marked demyelination and axonal loss. As a result, symptoms such as fatigue, numbness, weakness, depression, walking difficulties and spasticity frequently appear.

Although there is no cure for MS, several disease-modifying therapies are available. These can potentially slow the progression of disabilities and reduce the overall disease burden. This is of great interest from both an individual perspective, where increased disability is associated with a lowered health-related quality of life, and from a societal perspective, where increased disability is associated with larger costs.

Over the past decades exercise has been shown to be safe, tolerable and beneficial in persons with MS (PwMS). Hence, it is known to be an effective way of treating symptoms such as fatigue7, muscle weakness, walking impairments and depression. As with other chronic diseases, exercise for PwMS has been proposed as "medicine". However, in order to benefit from the positive effects of any kind of treatment (i.e. most medical drugs or exercise) one has to adhere to the prescriptions of the treatment (i.e. dose and timing). Despite all the potential benefits of exercise therapy for PwMS, one of the major challenges relate to long-term maintenance of exercise efforts.

An emerging concept that may hold the potential to increase the sustainability of exercise therapy is supervised "exercise booster sessions" (i.e. training sessions provided regularly throughout the follow-up period, to sustain effects of the preceding exercise intervention). These can be placed regularly during the follow-up period, where patients attend a number of supervised high-intensity exercise sessions, hereby trying to boost the effects of the preceding exercise intervention. Furthermore, exercise booster sessions can potentially motivate the patient to keep exercising throughout the follow up period.

However, the optimal way of utilizing this concept is still not fully understood, and has not yet been tried in neurological patients.

Therefore, the main purpose of the present study is to investigate how exercise booster sessions combined with usual care performed over a period of 40 weeks affects the sustainability of effects on functional capacity induced by a 12-week exercise intervention.

It is hypothesized that participants receiving exercise booster sessions + usual care during follow up will have a better functional capacity at follow up, than the participants receiving usual care only.

The study will be a randomized, multi-site, controlled trial. Participants will from the beginning be allocated to either aerobic training group, resistance training group or control group. After a 12 week exercise intervention, the exercise groups will be additionally randomized to receive either exercise booster sessions + standard care or just standard care in the 40 week follow up period.

The 12 week exercise intervention will consist of 2-3 weekly supervised exercise sessions. The training will be planned by exercise physiologists and performed in a progressive manner. To allow handling of a large number of participants, who is also geographically spread, the exercise intervention will be locally anchored, but at the same time supervised by student employees and controlled by internet- and telephonic communication.

Participants allocated to exercise booster sessions will receive two sessions every fifth week during the follow up period.

The power calculation is based on the primary purpose of the study which is to investigate the effect of frequently applied exercise booster sessions. To set the estimated number of participants, a two-sample two-sided power calculation has been conducted. Based on previous studies, a mean difference on functional capacity between the group receiving usual care and the group receiving exercise booster sessions + usual care, regardless of exercise intervention, is expected to be 6% with a standard deviation (SD) of ±10%.

The level of significance was set as 5% and a statistical power of 80%. According to the power calculation each group shall contain 60 participants (expected drop-out rate of 30 % is included).

The results of these studies can have great clinical implications in many ways. If we find that by adding exercise booster sessions in a follow up period, one can maintain, or maybe even improve, functional capacity over a long period, this would be a novel finding making ground for new rehabilitation opportunities

ELIGIBILITY:
Inclusion Criteria:

* A definite diagnosis of MS, according to the McDonald criteria
* Walking <650m on 6MWT.
* Exercising ≤ two sessions per week of moderate-to-high intensity during the past six months.

Exclusion Criteria:

* Comprise comorbidities (cardiovascular-, respiratory-, orthopedic- or other neurological diseases.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Change in functional capacity measured as a composite score of the six minute walk test and the 5x sit to stand test (5STS). | Baseline,12 weeks and 52 weeks.
  The six minute walk test it the distance covered during a six-minute maximal walking test. The 5STS is the time used to stand up from a chair and sit again five times.

SECONDARY OUTCOMES:
Change in functional capacity measured by the Six spot step test (SSST) | Baseline, 12 weeks and 52 weeks.
  SSST is a measure of walking ability, balance and coordination. Measured as the time to complete the six-spot course.
Change in functional capacity measured by the Multiple Sclerosis Functional Composite (MSFC) | Baseline, 12 weeks and 52 weeks.
  Composite score from Timed 25-Feet Walk Test (T25FWT), 9-Hole Peg Test (9HPT), Paced Auditory Serial Addition Test (PASAT)

OTHER OUTCOMES:
Change in physical activity, accelerometry | Baseline, 12 weeks and 52 weeks.
  Measurement of level of physical activity by wearing a accelerometer for 7 days at each time point. Measured in counts/min.
Change in aerobic capacity | Baseline, 12 weeks and 52 weeks.
  Maximal oxygen uptake test on bike ergometer, measured by indirect calorimetry.
Change in Multiple Sclerosis Walking Scale 12 (MSWS-12) | Baseline, 12 weeks and 52 weeks.
  Questionnaire assessing the impact of the disease on walking. Each question is scored from 1-5 and then summed and transformed to a 0-100 scale. Higher scores indicate a greater impact on walking.
Change in Modified Fatigue Impact Scale (MFIS) | Baseline, 12 weeks and 52 weeks.
  Questionnaire assessing the effects of fatigue on physical, cognitive and psychosocial functioning. The score of the MFIS is the sum of the scores for the 21 items. A higher score represents a higher impact of fatigue, in general or in relation to one of the above mentioned areas.
Change in Short Form Health Survey 36 (SF-36) | Baseline, 12 weeks and 52 weeks.
  Questionnaire assessing health status. The SF-36 consists of eight subscales, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Change in Hospital anxiety and depression scale (HADS) | Baseline, 12 weeks and 52 weeks.
  Questionnaire assessing anxiety and depression. It consists of two subscales (anxiety and depression), and should be scored separately. A higher score indicates a higher degree of anxiety and depression.
Change in self reported physical activity measured by the Baecke questionnaire. | Baseline, 12 weeks and 52 weeks.
  Questionnaire assessing the self reported amount of physical activity. This questionnaire quantifies the habitual physical activity level in three indexes: occupational (at work), sport (structured exercise) and leisure (leisure time). Each index is scored from 1 to 5, with 5 indicating the highest level of physical activity
Change in maximal strength | Baseline, 12 weeks and 52 weeks.
  Maximal strength measurement measured in the knee extensors by isokinetic dynamometry.
Change in functional capacity measured by the Timed Up and Go | Baseline, 12 weeks and 52 weeks
  The Timed up and Go is a test that evaluates functional components of mobility
Change in cognition measured by the SDMT | Baseline, 12 weeks and 52 weeks.
  The SDMT is a test measuring processing speed
Change in EQ-5D-5L | Baseline, 12 weeks and 52 weeks
  The EQ-5D-5L measures health related quality of life, and is measured both by a VAS scale and an index score
Change in societal costs measured by the HUQ | Baseline, 12 weeks and 52 weeks.
  The HUQ measures health utilization by assessing healthcare and medicine usage, and productivity.
Change in societal costs measured by the IPCQ. | Baseline, 12 weeks and 52 weeks.
  The IPCQ measures health utilization by assessing healthcare and medicine usage, and productivity.
Change in falls and fear of falling by the Falls Efficacy Scale | Baseline, 12 weeks and 52 weeks.
  The Falls Efficacy scale measures the concern participants have of falling

CONTACTS AND LOCATIONS:
Overall Officials: Laurits Taul-Madsen, MSc., Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All data will be stored in The Danish National Archives after completion of the project, and data can be accessed through request to The Danish National Archives.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after completion of the project, expectedly May 2024. The Danish National Archives stores data without a time frame (forever).
Access Criteria: Sharing of data can happen upon request to The Danish National Archives.

REFERENCES:
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Calabresi PA. Diagnosis and management of multiple sclerosis. Am Fam Physician. 2004 Nov 15;70(10):1935-44. PMID 15571060
- [Result] Pilutti LA, Platta ME, Motl RW, Latimer-Cheung AE. The safety of exercise training in multiple sclerosis: a systematic review. J Neurol Sci. 2014 Aug 15;343(1-2):3-7. doi: 10.1016/j.jns.2014.05.016. Epub 2014 May 15. PMID 24880538
- [Result] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Result] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Result] Heesen C, Bruce J, Gearing R, Moss-Morris R, Weinmann J, Hamalainen P, Motl R, Dalgas U, Kos D, Visioli F, Feys P, Solari A, Finlayson M, Eliasson L, Matthews V, Bogossian A, Liethmann K, Kopke S, Bissell P. Adherence to behavioural interventions in multiple sclerosis: Follow-up meeting report (AD@MS-2). Mult Scler J Exp Transl Clin. 2015 May 12;1:2055217315585333. doi: 10.1177/2055217315585333. eCollection 2015 Jan-Dec. PMID 28607693
- [Result] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Resistance training improves muscle strength and functional capacity in multiple sclerosis. Neurology. 2009 Nov 3;73(18):1478-84. doi: 10.1212/WNL.0b013e3181bf98b4. PMID 19884575
- [Result] Collett J, Dawes H, Meaney A, Sackley C, Barker K, Wade D, Izardi H, Bateman J, Duda J, Buckingham E. Exercise for multiple sclerosis: a single-blind randomized trial comparing three exercise intensities. Mult Scler. 2011 May;17(5):594-603. doi: 10.1177/1352458510391836. Epub 2011 Jan 19. PMID 21247971
- [Result] Kjolhede T, Vissing K, de Place L, Pedersen BG, Ringgaard S, Stenager E, Petersen T, Dalgas U. Neuromuscular adaptations to long-term progressive resistance training translates to improved functional capacity for people with multiple sclerosis and is maintained at follow-up. Mult Scler. 2015 Apr;21(5):599-611. doi: 10.1177/1352458514549402. Epub 2014 Sep 25. PMID 25257612
- [Derived] Taul-Madsen L, Hvid LG, Riis H, Brolos MK, Lundbye-Jensen J, Dalgas U. A head-to-head comparison of the effects of aerobic versus resistance training on physical capacity and physical function in people with multiple sclerosis: Results from the MSBOOST trial. Mult Scler. 2025 Feb;31(2):174-183. doi: 10.1177/13524585241305496. Epub 2024 Dec 30. PMID 39891566
- [Derived] Taul-Madsen L, Hvid LG, Sellebjerg F, Christensen JR, Ratzer R, Sejbaek T, Svendsen KB, Papp V, Hojsgaard Chow H, Lundbye-Jensen J, Dawes H, Dalgas U. Study protocol: effects of exercise booster sessions on preservation of exercise-induced adaptations in persons with multiple sclerosis, a multicentre randomised controlled trial-the MS BOOSTER trial. BMJ Open. 2024 Aug 17;14(8):e085241. doi: 10.1136/bmjopen-2024-085241. PMID 39153792